CLINICAL TRIAL: NCT01134419
Title: Implementing a Comprehensive Handoff Program to Improve Pediatric Patient Safety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: Harvard Risk Management Foundation (Other)
Responsible Party: Principal Investigator, Christopher Landrigan, Research and Fellowship Director, Inpatient Pediatrics Service, Boston Children's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: X09-01-0040
Record Dates: First submitted 2010-05-25; First posted 2010-06-02 (Estimated); Last update posted 2013-05-16 (Estimated); Status verified 2013-05

CONDITIONS: Patient Safety; Resident Workflow; Resident Experience
Keywords: Patient Safety; Medical Errors; Handoff; Sign-out; Resident; Intern; Graduate Medical Education

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Computerized Handoff Tool plus training (Experimental): Computerized handoff tool implemented together with team training for residents
  Interventions: Other: Computerized handoff tool; Other: Team training
- Team training only (Active Comparator): No computerized tool
  Interventions: Other: Team training

INTERVENTIONS:
Other: Computerized handoff tool — Informatics tool to aid in transfer of patient care information
  Arms: Computerized Handoff Tool plus training
Other: Team training — Teamwork training and revisions of handoff structure to optimize teamwork skills and verbal communications

SUMMARY:
The investigators propose to test the hypothesis that implementation of a comprehensive handoff program (CHP) - i.e., implementation of a computerized handoff tool along with teamwork training for pediatric residents on inpatient units at Children's Hospital Boston - will lead to reductions in resident miscommunications / medical errors and improvements in workflow and experience on the wards.

DETAILED DESCRIPTION:
Following collection of baseline data on two inpatient pediatric wards, teamwork training is to be provided to all pediatric residents. On our primary intervention unit, this will be accompanied by the introduction of a new computerized handoff tool that facilitates accurate transmission of data. The effects of this combined intervention on safety and workflow will be assessed on the primary intervention ward as compared with the historical control unit and the concurrent unit that received teamwork training without the computerized tool.

ELIGIBILITY:
Inclusion Criteria:

* all residents working on study units during study period, except as below

Exclusion Criteria:

* residents on the teamwork only unit who have previously been on the primary intervention unit

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2009-07; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Rates of resident-related communication and total medical errors | July 2010
  Resident-related medical errors (including medication-related, diagnostic, and procedural) detected using a multi-pronged prospective surveillance methodology that involves 5d/week chart review, review of hospital incident reports, and collection of staff reports. Resident-related defined as involving a resident research subject. Communication errors are those medical errors attributable to communication failures.

SECONDARY OUTCOMES:
Rates of total medical errors | July 2010
  As above, but includes both those errors involving residents and those involving all other clinical personnel.
Minutes residents spend updating the signout; minutes spent in direct patient care; minutes spent working at computer | July 2010
Resident reported experience of care | July 2010
  Self-reported, Likert scales on survey instruments.
Rates of verbal miscommunications | July 2010
  Detected by direct observation, audio recording, then rating using study instrument developed for this purpose.
Rates of written miscommunications | July 2010
  Detected by detailed review of written signouts, rated using study instrument developed for this purpose.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher P Landrigan, MD, MPH, Principal Investigator — Boston Children's Hospital
Locations (1):
- Children's Hospital Boston, Boston, Massachusetts, United States